CLINICAL TRIAL: NCT02850497
Title: 6-month Intracoronary Optical Coherence Tomography (OCT) Evaluation of Endothelization and Malapposition of Three New Generation Drug Eluting Stent: CRE8, Biomatrix and Xience
Brief Title: 6-month Intracoronary Optical Coherence Tomography (OCT) Evaluation of Three New Generation Drug Eluting Stent
Acronym: CREBX-OCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Cristina Giglioli, MD, MD, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 875/13
Record Dates: First submitted 2015-04-30; First posted 2016-08-01 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Recurrent Angina After Coronary Stent Placement
Keywords: optical coherence tomography; malapposition; endothelization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CRE8 stent (Active Comparator): Treatment with CRE8 stent implantation and evaluated with optical coherence tomography at 6 months
  Interventions: Device: optical coherence tomography at 6 months
- Biomatrix stent (Active Comparator): Treatment with Biomatrix stent implantation and evaluated with optical coherence tomography at 6 months
  Interventions: Device: optical coherence tomography at 6 months
- patients treated with Xience stent (Active Comparator): Treatment with Xience stent implantation and evaluated with optical coherence tomography at 6 months
  Interventions: Device: optical coherence tomography at 6 months

INTERVENTIONS:
Device: optical coherence tomography at 6 months — 6-month evaluation of malapposition and endothelization with the use of intracoronary optical coherence tomography

SUMMARY:
Aim of this study is to compare at 6 months follow-up, endothelization and malapposition, evaluated by means of optical coherence tomography, in terms of number of struts not endothelized or malapposed, after the implantation of three new generation stent: Cre8, Biomatrix and Xience.

DETAILED DESCRIPTION:
This is a randomized study aimed at evaluating in 60 patients with either acute coronary syndromes or stable coronary artery disease submitted with PCI and stenting, endothelization and malapposition at 6 months follow-up (primary endpoint), evaluated by means of optical coherence tomography in terms of number of struts not re-endothelized or malapposed, after the implantation of three new generation stent: Cre8, Biomatrix and Xience. Further clinical follow-up will be performed to evaluate MACE at 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with stable angina or acute coronary syndromes submitted to coronary angioplasty on a coronary with a vessel diameter > 2,5 mm

Exclusion Criteria:

* Known allergy to antithrombotic drugs or to other components of the stent studied Planned surgery 6 months within angioplasty

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
stent struts coverage assessed by means of intracoronary optical coherence tomography | 6 months

SECONDARY OUTCOMES:
MACE (cardiovascular death, myocardial infarction, stroke and target vessel revascularization) | 12 months
inducible ischemia at myocardial scintigraphy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Giglioli, MD, Principal Investigator — Azienda Ospedaliero-Universitaria Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided
To date a decision has not been taken with regard to a possible plan to share data

REFERENCES:
- [Derived] Giglioli C, Formentini C, Romano SM, Cecchi E, Baldereschi GJ, Landi D, Chiostri M, Prati F, Marchionni N. Vulnerable struts with CRE8, Biomatrix and Xience stents assessed with OCT and their correlation with clinical variables at 6-month follow-up: the CREBX-OCT study. Int J Cardiovasc Imaging. 2020 Feb;36(2):217-230. doi: 10.1007/s10554-019-01719-1. Epub 2019 Oct 30. PMID 31667661